CLINICAL TRIAL: NCT05023603
Title: Social Determinants of Health and Cognitive Factors in Carpal Tunnel Syndrome
Brief Title: Social and Cognitive Factors in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Hospital Clínico La Florida (Other)
Responsible Party: Principal Investigator, Rodrigo Ignacio Nunez Cortes, Principal Investigator, Hospital Clínico La Florida
Other Study IDs: RNC0032018
Record Dates: First submitted 2021-08-22; First posted 2021-08-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Carpal Tunnel Syndrome; Carpal Tunnel
Keywords: Chronic pain; Disability; psychosocial factors; social determinants of health
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: self-report questionnaire — Individual subject factors included and self-report questionnaires will be collected through an interview process.
  Other Names: data collection only

SUMMARY:
Carpal tunnel syndrome (CTS) is a compressive peripheral neuropathy, characterized by pain, tingling sensation and paresthesia in the territory of the median nerve, symptoms modulated by psychosocial factors (eg, catastrophic thinking, depression, anxiety).

The objective of the study is to determine those psychological and social components that influence the symptoms and function of patients with CTS.

An observational cross-sectional design will be performed in patients with CTS. The patients will be selected consecutively in two hospitals of the South East Metropolitan Health Service (Santiago, Chile). The study variables will include: Perception of pain using the Visual Analogue Scale (VAS), the extent of symptoms will be evaluated using the Katz diagram; Functional assessment using the abbreviated version of the Disabilities of the Arm, Shoulder and Hand Questionnaire (QuickDASH); Catastrophic thinking as a response to pain using the Pain Catastrophizing Scale (PCS), fear of movement using the Tampa Scale for Kinesiophobia (TSK-11), and emotional state was assessed using the Hospital Anxiety and Depression Scale (HADS). Both are valid and reliable measures used to evaluate the influence of psychosocial factors in patients with CTS. Individual subject factors including duration of symptoms, type of work (desk / non-desk), BMI, age, gender, educational level and economic income will be collected through an interview process.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, moderate or severe CTS medical diagnosis, duration of symptoms for more than three months, acceptance to participate in the study.

Exclusion Criteria:

* Inability to understand instructions, non-controlled mental health pathology, cognitive problems, and previous surgery in the upper limb.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Carpal tunnel syndrome (CTS) is a compressive peripheral neuropathy, characterized by pain, a tingling sensation and paraesthesia over the skin territory of the median nerve.
  The patient's medical history, the presence of risk factors, and the characteristics of the symptoms are key aspects for establishing a suitable differential diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | Baseline (0 weeks)
  Pain will be measured by the Visual Analog Scale for pain (VAS) from 0 to 10, where higher values represent a worse outcome.
Disability in upper-limb | Baseline (0 weeks)
  The Perception of patients of their disability in upper-limb evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH) Spanish version Outcome Measure is a 30-item scored 1-5 (referencia). The assigned values for all completed responses are simply summed and averaged. Scoring: The assigned values for all completed responses are simply summed and averaged and higher values represent a worse Disability in upper-limb
Hand diagrams | Baseline (0 weeks)
  To define total area marked for pain and numbness. The areas of the hand are marked by the patient and the marked area is quantified in square centimeters.

SECONDARY OUTCOMES:
Pain Interference: Kinesiophobia | Baseline (0 weeks)
  Kinesiophobia will be evaluated by Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz-Párraga, 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
Emotional status: Hospital Anxiety and Depression Scale (HAD). | Baseline (0 weeks)
  Patient's emotional state will be evaluated by Hospital Anxiety and Depression Scale (HAD), which assess the level of anxiety and depression. Subscales and score range are Anxiety (0-21) and Depression (0-21). Scoring: items of each subscale are summed, indicating: 0-7 normality, 8-10 probably case, 11-21 anxiety or depression clinical case. Higher values represent a worse outcome.
Pain Catastrophizing Scale (PCS) | Baseline (0 weeks)
  To assess catastrophic thinking as a response to pain through 13 statements with 4 possible options from 1 "not at all" to 4 "all the time". a higher score indicates a higher catastrophic thinking
Educational level | Baseline (0 weeks)
  At an educational level, it will be categorized according to: complete primary education, complete secondary education and completed university studies.
Grip strength | Baseline (0 weeks)
  Measured using a Jamar dynamometer (Preston, Clifton, NJ) in the second handle position, following the recommendations of the American Society of Hand Therapists
Lateral pinch strength | Baseline (0 weeks)
  Measured using a pinch meter (Preston, Clifton, NJ), following the recommendations of the American Society of Hand Therapists
Socioeconomic status | Baseline (0 weeks)
  This indicator is calculated by dividing the effective income of each family by its index of needs. Effective income: monthly average of income received, including work, capital and pensions.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Hospital Provincia Cordillera, Santiago
  - Hospital Clínico la Florida, Santiago

IPD SHARING:
Plan to Share IPD: Undecided